CLINICAL TRIAL: NCT00002230
Title: A Randomized, Placebo-Controlled Study of the Safety and Efficacy of Efavirenz, Didanosine, and Stavudine in Combination With or Without Hydroxyurea in Antiretroviral Naive or Experienced HIV-Infected Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Northwestern University (Other)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 296A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-06

CONDITIONS: HIV Infections
Keywords: Didanosine; Drug Therapy, Combination; Stavudine; Hydroxyurea; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections | interventions — Hydroxyurea; efavirenz; Stavudine; Didanosine

INTERVENTIONS:
Drug: Hydroxyurea
Drug: Efavirenz
Drug: Stavudine
Drug: Didanosine

SUMMARY:
To determine the virologic benefits associated with the addition of hydroxyurea (HU) to combination drug therapy with didanosine (ddI), stavudine (d4T), and efavirenz (DMP) in HIV-infected patients. To assess the safety and tolerance of this regimen, with or without HU.

DETAILED DESCRIPTION:
HU or placebo is added 30-60 days after the initiation of DMP, ddI, and d4T combination therapy. Patients are stratified according to antiretroviral experience (naive or experienced). Patients are followed for 48 weeks to determine safety, efficacy, and effect of treatment on viral, immunologic,and biochemical parameters.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV infection, as documented by a licensed ELISA that is confirmed either by Western blot, positive HIV culture, positive HIV antigen, positive plasma HIV RNA, or a second antibody test positive by a method other than ELISA.
* CD4 cell count of at least 100 cells/mm3 within 30 days of study entry.
* Over 500 HIV-1 RNA copies/ml as measured by the Roche Amplicor or Ultra Sensitive Assay within 30 days of study entry.
* Treatment-experienced patients must have documented HIV RNA values of less than or equal to 100,000 copies/ml within 30 days of study entry.

Prior Treatment:

Excluded:

Acute therapy for an infection or other medical illness. Acute therapy must have been completed 14 days prior to the time of study entry.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

Malignancy requiring systemic therapy.

Patients with the following prior conditions are excluded:

* History of acute or chronic pancreatitis.
* History of generalized peripheral neuropathy.
* Inability to tolerate ddI at 200-400 mg/day or d4T at 60-80 mg/day. For purposes of this study, intolerance will be defined as the same recurrent toxicities requiring dose interruptions and dose reductions or permanent discontinuation of the drugs (other than Grade 3 or 4 anemia).

Prior Medication:

Excluded:

Antiretroviral therapy. If antiretroviral-experienced, no prior NNRTI's or HU and no more than 12 weeks experience with ddI and/or d4T. Protease inhibitor experience is allowed. Experienced patients must be on a stable antiretroviral therapy 30 days prior to study screening and continue this regimen until study entry.

Risk Behavior:

Excluded:

Current ethanol abuse by personal history or a report from a primary physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100

CONTACTS AND LOCATIONS:
Overall Officials: Robert Murphy, Study Chair
Locations (1):
- Northwestern Univ Med School, Chicago, Illinois, United States